CLINICAL TRIAL: NCT05225597
Title: The Effect of Intracameral Carbachol and Epinephrine Use on Choroidal Thickness After Uncomplicated Phacoemulsification
Brief Title: The Effect of Intracameral Carbachol and Epinephrine on Choroidal Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hasan Burhanettin Kapti, Principal Investigator, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PANTONE 287 C
Record Dates: First submitted 2022-01-14; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Epinephrine Toxicity; Cataract; Carbachol Adverse Reaction; Choroid Disease
Keywords: choroidal thickness; carbachol; epinephrine; phacoemulsification; optical coherence tomography
MeSH Terms: conditions — Cataract; Choroid Diseases

STUDY DESIGN:
Intervention Model Description: This study consisted of three groups: epinephrine group, carbachol group, and control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were unaware of the group in which they were assigned. The person evaluating the results did not know which result belonged to which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- epinephrine (Active Comparator): In the epinephrine group, 0.2 mL of epinephrine (1:5000 solution) was used immediately after making the clear corneal incision during cataract surgery
  Interventions: Procedure: Intracameral administration of epinephrine and carbachol during cataract surgery
- carbachol (Active Comparator): In the carbachol group, a 0.5 ml dose of 0.01% carbachol solution (Miostat®, Alcon Laboratories, Inc., Fort Worth, TX) was given intracamerally immediately after viscoelastic matter removal following IOL implantation
  Interventions: Procedure: Intracameral administration of epinephrine and carbachol during cataract surgery
- control (No Intervention): The control group was given neither epinephrine nor carbachol. Standard cataract surgery was performed

INTERVENTIONS:
Procedure: Intracameral administration of epinephrine and carbachol during cataract surgery — All surgeries were performed by the same surgeon using a similar technique, under topical anesthesia (0.05% proparacaine HCL), and with a 2.8 mm temporal clear corneal incision. After making the incision, 0.2 mL of preservative-free epinephrine (1:5000) was injected into the epinephrine group only. After complete hydrodissection, the nucleus was removed using the stop and chop technique. Phacoemulsification time (range: 30-60 s) was similar in all patients, while the phacoemulsification strength was set to 35%-40% for all operations. The cortex was aspirated. Before implanting a one-piece foldable hydrophobic acrylic intraocular lens (IOL) into the capsular bag, 1% sodium hyaluronate (ophthalmic viscosurgical device, Healon) was injected into the capsular bag. After removal of the viscoelastic material, only the carbachol group was given 0.5 ml of 0.01% carbachol solution intracamerally. Hydration with balanced salt solution was used to close the corneal incisions.
  Arms: carbachol; epinephrine

SUMMARY:
81 eyes of 81 patients undergoing cataract surgery were included in this prospective interventional study. During cataract surgery, intracameral carbachol was applied to 27 eyes, intracameral epinephrine was administered to 20 eyes and 34 eyes were the control group. Macular choroidal thickness measurement was performed before, 1 day, and 1 week after phacoemulsification surgery in all patients using optical coherence tomography.

DETAILED DESCRIPTION:
This study consisted of three groups: epinephrine group, carbachol group, and control group. Intracameral carbachol and epinephrine was not used for complication management. In the epinephrine group, 0.2 mL of epinephrine (1:5000 solution) was used immediately after making the clear corneal incision. In the carbachol group, a 0.5 ml dose of 0.01% carbachol solution (Miostat®, Alcon Laboratories, Inc., Fort Worth, TX) was given intracamerally immediately after viscoelastic matter removal following IOL implantation. The control group was given neither epinephrine nor carbachol.

Mydriasis was induced using combined 2.5% phenylephrine and 1.0% tropicamide topical drops before surgery. All surgeries were performed by the same surgeon (HBK) using a similar technique, under topical anesthesia (0.05% proparacaine HCL), and with a 2.8 mm temporal clear corneal incision. After making the incision, 0.2 mL of preservative-free epinephrine (1:5000) was injected into the epinephrine group only. A combination of 1.6% sodium hyaluronate and 4% chondroitin sulfate (ophthalmic viscosurgical device, Discovisc, Alcon Laboratories, Inc.) was used during capsulorhexis in all three groups, and Alcon Infiniti System (Alcon Laboratories Inc.) was used for phacoemulsification. A continuous curvilinear capsulorhexis of 4.5-5.5 mm was created. After complete hydrodissection, the nucleus was removed using the stop and chop technique. Phacoemulsification time (range: 30-60 s) was similar in all patients, while the phacoemulsification strength was set to 35%-40% for all operations. The cortex was aspirated in irrigation/aspiration mode. Before implanting a one-piece foldable hydrophobic acrylic IOL into the capsular bag, 1% sodium hyaluronate (ophthalmic viscosurgical device, Healon) was injected into the capsular bag. After removal of the viscoelastic material, only the carbachol group was given 0.5 ml of 0.01% carbachol solution intracamerally. Hydration with balanced salt solution was used to close the corneal incisions. Topical moxifloxacin, nepafenac, and prednisolone acetate eye drops were given to all patients six times a day for the first week. Prednisolone acetate was then reduced and discontinued 4 weeks after the operation.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* patients with cataracts

Exclusion Criteria:

* hypertension and diabetes
* ocular problems such as uveitis, glaucoma, amblyopia
* maculopathy, retinal dystrophy
* any previous ocular surgery
* eye trauma
* congenital cataracts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
choroidal thickness(CT) | preoperatively, on postoperative day 1, and in postoperative week 1
  CT measurement was performed using a Cirrus HD(high definition) 500 spectral OCT (optical coherence tomography) platform (Carl Zeiss Meditec, Dublin, California, USA). Subfoveal, nasal, temporal, lower choroidal thickness, and upper choroidal thickness were measured manually by two blinded observers with 0.5-mm intervals in vertical and horizontal sections having a length of 4 mm. The distance between the outer hyper-reflective border of the retinal pigment epithelium and the inner scleral surface was considered. Average data obtained by two observers were used in statistical analysis.

SECONDARY OUTCOMES:
intraocular pressure | before, 1 day, and 1 week after surgery
  Intraocular pressure was measured in all patients using a non-contact tonometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan B Kaptı, MD, Principal Investigator — Ordu University
Locations (1):
- Ordu University, Ordu, ABD Dışında, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No